CLINICAL TRIAL: NCT04832971
Title: A Double-blind, Placebo-controlled Phase 2b Study to Evaluate the Efficacy and Safety of ARO-ANG3 in Adults With Mixed Dyslipidemia
Brief Title: Study of ARO-ANG3 in Adults With Mixed Dyslipidemia
Acronym: ARCHES-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AROANG3-2001
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Mixed Dyslipidemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ARO-ANG3 50 mg (Experimental): Two doses of ARO-ANG3 by subcutaneous (sc) injection at Day 1 and Week 12 during double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
  Interventions: Drug: ARO-ANG3
- ARO-ANG3 100 mg (Experimental): Two doses of ARO-ANG3 bysc injection at Day 1 and Week 12 during double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
  Interventions: Drug: ARO-ANG3
- ARO-ANG3 200 mg (Experimental): Two doses of ARO-ANG3 by sc injection at Day 1 and Week 12 during double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
  Interventions: Drug: ARO-ANG3
- Placebo (Placebo Comparator): Calculated volume to match active treatment by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
  Interventions: Drug: ARO-ANG3; Drug: Placebo

INTERVENTIONS:
Drug: ARO-ANG3 — ARO-ANG3 Injection
Drug: Placebo — Sterile Normal Saline (0.9% NaCl)
  Arms: Placebo

SUMMARY:
The purpose of AROANG3-2001 is to evaluate the efficacy and safety of ARO-ANG3 in participants with mixed dyslipidemia. Participants will initially receive 2 subcutaneous injections of ARO-ANG3 or placebo. Participants who complete the double-blind treatment period may opt to continue in an open-label extension during which they will receive up to 8 doses of ARO-ANG3.

ELIGIBILITY:
Inclusion Criteria:

* Based on medical history, evidence of triglycerides (TG) ≥ 150 mg/dL but ≤ 499 mg/dL
* Fasting levels at Screening of LDL-C ≥ 70 mg/dL OR non-HDL-C ≥ 100 mg/dL after at least 4 weeks of stable diet and stable optimal statin therapy
* Mean fasting TG ≥ 150 mg/dL and ≤ 499 mg/dL during Screening collected at two separate and consecutive visits and at least 7 days apart and not more than 17 days apart
* Willing to follow diet counseling and maintain a stable diet per Investigator judgment based on local standard of care
* Participants of childbearing potential must agree to use highly-effective contraception during the study and for at least 24 weeks from last dose of study medication
* Women of childbearing potential must have a negative pregnancy test and cannot be breastfeeding
* Women of childbearing potential on hormonal contraceptives must be stable on the medication for ≥ 2 menstrual cycles prior to Day 1
* Men must not donate sperm during the study and for at least 24 weeks following the last dose of study medication
* Able and willing to provide written informed consent and to comply with study requirements

Exclusion Criteria:

* Current use or use within 365 days from Day 1 of any hepatocyte targeted siRNA or antisense oligonucleotide molecule
* Active pancreatitis within 12 weeks prior to Day 1
* Any planned bariatric surgery or similar procedures to induce weight loss from consent to end of study
* Acute coronary syndrome event within 24 weeks of Day 1
* Major surgery within 12 weeks of Day 1 or planned surgery during the study
* Planned coronary intervention (e.g., stent placement or heart bypass) during the study
* Uncontrolled hypertension
* Human immunodeficiency virus (HIV) infection, seropositive for Hepatitis B (HBV), seropositive for Hepatitis C (HCV)
* Uncontrolled hypothyroidism or hyperthyroidism
* Hemorrhagic stroke within 24 weeks of Day 1
* History of bleeding diathesis or coagulopathy
* Current diagnosis of nephrotic syndrome
* Systemic use of corticosteroids or anabolic steroids within 4 weeks prior to Day 1 or planned use during the study
* Malignancy within the last 2 years prior to date of consent requiring systemic treatment (some exceptions apply)

Note: additional inclusion/exclusion criteria may apply per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (13):
  - Research Site 5, Huntington Park, California
  - Research Site 7, Hialeah, Florida
  - Research Site 17, Miami, Florida
  - Research Site 8, Port Orange, Florida
  - Research Site 24, Minneapolis, Minnesota
  - Research Site 10, Omaha, Nebraska
  - Research Site 23, Las Vegas, Nevada
  - Research Site 22, New York, New York
  - Research Site 15, Greensboro, North Carolina
  - Research Site 2, Morehead City, North Carolina
  - Research Site 1, Marion, Ohio
  - Research Site 4, Camp Hill, Pennsylvania
  - Research Site 11, Houston, Texas
- Australia (3):
  - Research Site 6, Blacktown, New South Wales
  - Research Site 21, Sippy Downs, Queensland
  - Research Site 18, Nedlands
- Canada (4):
  - Research Site 25, London, Ontario
  - Research Site 16, Chicoutimi, Quebec
  - Research Site 12, Québec
  - Research Site 9, Québec
- New Zealand (4):
  - Research Site 19, Birkenhead
  - Research Site 13, Christchurch
  - Research Site 20, Hamilton
  - Research Site 14, Rotorua

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenson RS, Gaudet D, Hegele RA, Ballantyne CM, Nicholls SJ, Lucas KJ, San Martin J, Zhou R, Muhsin M, Chang T, Hellawell J, Watts GF; ARCHES-2 Trial Team. Zodasiran, an RNAi Therapeutic Targeting ANGPTL3, for Mixed Hyperlipidemia. N Engl J Med. 2024 Sep 12;391(10):913-925. doi: 10.1056/NEJMoa2404147. Epub 2024 May 29. PMID 38809174
- [Derived] Dimitriadis K, Theofilis P, Iliakis P, Pyrpyris N, Dri E, Sakalidis A, Soulaidopoulos S, Tsioufis P, Fragkoulis C, Chrysohoou C, Tsiachris D, Tsioufis K. Management of dyslipidemia in coronary artery disease: the present and the future. Coron Artery Dis. 2024 Sep 1;35(6):516-524. doi: 10.1097/MCA.0000000000001375. Epub 2024 Apr 29. PMID 38682459

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo calculated volume to match active treatment by subcutaneous (sc) injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- ARO-ANG3 50 mg: ARO-ANG3 50 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- ARO-ANG3 100 mg: ARO-ANG3 100 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- ARO-ANG3 200 mg: ARO-ANG3 200 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- Placebo/ARO-ANG3 50 mg: Placebo calculated volume to match active treatment by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 50 mg by sc injection during the open-label extension period.
- ARO-ANG3 50 mg/ARO-ANG3 50 mg: ARO-ANG3 50 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 50 mg by sc injection during the open-label extension period.
- Placebo/ARO-ANG3 100 mg: Placebo calculated volume to match active treatment by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 100 mg by sc injection during the open-label extension period.
- ARO-ANG3 100 mg/ARO-ANG3 100 mg: ARO-ANG3 100 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 100 mg by sc injection during the open-label extension period.
- Placebo/ARO-ANG3 200 mg: Placebo calculated volume to match active treatment by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 200 mg by sc injection during the open-label extension period.
- ARO-ANG3 200mg/ARO-ANG3 200mg: ARO-ANG3 200 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 200 mg by sc injection during the open-label extension period.
Period: Double-Blind (DB) Treatment Period
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Started | 51 | 51 | 51 | 51 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed Double-Blind (DB) Treatment Period) | 48 | 46 | 47 | 50 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other, Not Specified | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Extension (OLE) Period
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Started (Enrolled in OLE Treatment Period) | 0 | 0 | 0 | 0 | 13 | 36 | 14 | 39 | 13 | 41
Completed (Completed 24-month Treatment at OLE Treatment Period) | 0 | 0 | 0 | 0 | 5 | 17 | 3 | 14 | 6 | 17
Not Completed | 0 | 0 | 0 | 0 | 8 | 19 | 11 | 25 | 7 | 24
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 7 | 18 | 7 | 19 | 4 | 19
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 3
Not completed — Other, Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ARO-ANG3 100 mg: ARO-ANG3 100 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period.Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- Total: Total of all reporting groups
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg | Total
Number analyzed (Participants) | 51 | 51 | 51 | 51 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.30) | 60.4 (12.68) | 60.0 (9.89) | 61.5 (12.53) | 60.5 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 22 | 24 | 95
  Male | 27 | 26 | 29 | 27 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 18 | 13 | 55
  Not Hispanic or Latino | 39 | 39 | 33 | 38 | 149
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 49 | 49 | 49 | 195
  Black or African American | 1 | 1 | 1 | 0 | 3
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Other | 1 | 0 | 0 | 1 | 2
Mean Triglycerides (TG) at Baseline [Mean (Standard Deviation); unit: mg/dL] | 235.15 (86.117) | 242.47 (79.864) | 246.71 (97.996) | 259.97 (93.320) | 246.08 (89.386)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting TG at Week 24
Time Frame: Baseline, Week 24
Population: Full Analysis Set: All randomized participants who received at least 1 dose of investigational product (IP) during the study period, analyzed according to the treatment assigned at randomization.Observed cases.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Groups:
- Placebo: Placebo calculated volume to match active treatment by subcutaneous (sc) at Day 1 and Week 12 injection during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 47 | 47 | 47 | 49
percentage change | 7.55 (3.774) | -43.67 (3.770) | -49.01 (3.777) | -55.57 (3.726)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures (MMRM) — Model includes treatment arm, study visit, randomization stratification factor (LDL-C at Screening [≥100 mg/dL vs <100 mg/dL]),and baseline value as model terms. Model also includes treatment by visit and treatment by baseline as interaction terms; Difference vs. Placebo at Week 24 = -51.22, 95% CI 2-sided [-61.73 to -40.70] — ARO-ANG3 - Placebo
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p < .0001, Holm method — The adjusted p-value is calculated using the Holm method for multiplicity adjustment
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo at Week 24 = -56.56, 95% CI 2-sided [-67.09 to -46.04] — ARO-ANG3 - Placebo
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p < .0001, Holm method — The adjusted p-value is calculated using the Holm method for multiplicity adjustment
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Mixed Model with Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -63.11, 95% CI 2-sided [-73.56 to -52.66]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Holm method — The adjusted p-value is calculated using the Holm method for multiplicity adjustment

2. Secondary Outcome: Percent Change From Baseline in Fasting TG Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: Full Analysis Set: All randomized participants who received at least 1 dose of IP during the study period, analyzed according to the treatment assigned at randomization. Observed cases.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 51 | 50 | 48 | 50
  Week 4 | 7.00 (3.583) | -41.52 (3.604) | -52.22 (3.658) | -56.21 (3.619)
  Week 8: number analyzed (Participants) | 51 | 50 | 49 | 49
  Week 8 | 13.58 (4.188) | -41.01 (4.217) | -47.73 (4.250) | -52.55 (4.257)
  Week 12: number analyzed (Participants) | 47 | 48 | 48 | 51
  Week 12 | 2.17 (4.305) | -42.79 (4.269) | -41.71 (4.274) | -49.84 (4.183)
  Week 16: number analyzed (Participants) | 49 | 49 | 49 | 51
  Week 16 | 17.18 (6.952) | -48.48 (6.947) | -51.99 (6.942) | -58.73 (6.820)
  Week 20: number analyzed (Participants) | 48 | 48 | 48 | 51
  Week 20 | 11.54 (5.930) | -48.70 (5.928) | -52.73 (5.942) | -57.97 (5.790)
  Week 24: number analyzed (Participants) | 47 | 47 | 47 | 49
  Week 24 | 7.55 (3.774) | -43.67 (3.770) | -49.01 (3.777) | -55.57 (3.726)
  Week 28: number analyzed (Participants) | 48 | 47 | 45 | 49
  Week 28 | 7.24 (3.950) | -41.38 (3.966) | -43.95 (4.039) | -54.39 (3.920)
  Week 36: number analyzed (Participants) | 48 | 47 | 46 | 50
  Week 36 | -0.43 (3.798) | -34.49 (3.809) | -38.33 (3.850) | -51.63 (3.750)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — MMRM model includes treatment arm, study visit, randomization stratification factor (level of LDL-C at Screening [≥100 mg/dL versus <100 mg/dL]),and baseline value as model terms, and treatment by visit and treatment by baseline as interaction terms; Difference = -48.52, 95% CI 2-sided [-58.53 to -38.51]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -59.21, 95% CI 2-sided [-69.30 to -49.12]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -63.21, 95% CI 2-sided [-73.24 to -53.18]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p < .0001, m — [p-value comment as in outcome 2, analysis 1]; Difference = -54.60, 95% CI 2-sided [-66.31 to -42.89]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -61.31, 95% CI 2-sided [-73.07 to -49.55]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -66.13, 95% CI 2-sided [-77.90 to -54.37]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -44.96, 95% CI 2-sided [-56.91 to -33.01]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -43.87, 95% CI 2-sided [-55.83 to -31.92]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -52.00, 95% CI 2-sided [-63.83 to -40.18]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 50 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -65.66, 95% CI 2-sided [-85.04 to -46.29]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -69.17, 95% CI 2-sided [-88.54 to -49.80]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -75.91, 95% CI 2-sided [-95.11 to -56.71]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -60.24, 95% CI 2-sided [-76.78 to -43.71]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -64.27, 95% CI 2-sided [-80.83 to -47.72]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -69.52, 95% CI 2-sided [-85.85 to -53.18]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -51.22, 95% CI 2-sided [-61.73 to -40.70]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -56.56, 95% CI 2-sided [-67.09 to -46.04]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -63.11, 95% CI 2-sided [-73.56 to -52.66]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -48.62, 95% CI 2-sided [-59.66 to -37.59]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -51.19, 95% CI 2-sided [-62.32 to -40.05]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -61.63, 95% CI 2-sided [-72.60 to -50.67]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -34.06, 95% CI 2-sided [-44.65 to -23.46]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -37.90, 95% CI 2-sided [-48.56 to -27.25]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -51.19, 95% CI 2-sided [-61.71 to -40.68]

3. Secondary Outcome: Percent Change From Baseline in Fasting Non-High-Density Lipoprotein-Cholesterol (Non-HDL-C) at Week 24
Time Frame: Baseline, Week 24
Population: Full Analysis Set: All randomized participants who received at least 1 dose of IP during the study period, analyzed according to the treatment assigned at randomization.Observed cases.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 47 | 47 | 47 | 49
percentage change | 4.2 (3.31) | -25.1 (3.31) | -24.6 (3.31) | -32.2 (3.26)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -29.2, 95% CI 2-sided [-38.5 to -20.0]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -28.7, 95% CI 2-sided [-37.9 to -19.5]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -36.4, 95% CI 2-sided [-45.5 to -27.2]

4. Secondary Outcome: Percent Change From Baseline in Fasting Non-HDL-C Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Groups:
- Placebo: Placebo calculated volume to match active treatment by subcutaneous (sc) injection for Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 51 | 50 | 48 | 50
  Week 4 | 5.2 (2.51) | -23.5 (2.52) | -25.3 (2.55) | -32.9 (2.50)
  Week 8: number analyzed (Participants) | 51 | 50 | 49 | 49
  Week 8 | 3.7 (3.02) | -24.4 (3.04) | -22.8 (3.04) | -30.3 (3.02)
  Week 12: number analyzed (Participants) | 47 | 48 | 48 | 51
  Week 12 | 3.4 (3.06) | -22.8 (3.04) | -18.4 (3.04) | -28.1 (2.97)
  Week 16: number analyzed (Participants) | 49 | 49 | 49 | 51
  Week 16 | 2.5 (2.86) | -26.8 (2.86) | -28.3 (2.85) | -37.0 (2.81)
  Week 20: number analyzed (Participants) | 48 | 48 | 48 | 51
  Week 20 | 0.8 (2.71) | -28.1 (2.70) | -26.5 (2.69) | -34.1 (2.64)
  Week 24: number analyzed (Participants) | 47 | 47 | 47 | 49
  Week 24 | 4.2 (3.31) | -25.1 (3.31) | -24.6 (3.31) | -32.2 (3.26)
  Week 28: number analyzed (Participants) | 48 | 47 | 45 | 49
  Week 28 | 1.2 (3.00) | -23.1 (3.01) | -22.3 (3.04) | -30.0 (2.96)
  Week 36: number analyzed (Participants) | 48 | 47 | 46 | 50
  Week 36 | -1.5 (3.19) | -20.2 (3.21) | -17.3 (3.23) | -24.1 (3.14)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -28.7, 95% CI 2-sided [-35.7 to -21.7]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -30.5, 95% CI 2-sided [-37.5 to -23.4]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -38.1, 95% CI 2-sided [-45.1 to -31.2]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -28.2, 95% CI 2-sided [-36.6 to -19.7]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -26.6, 95% CI 2-sided [-35.0 to -18.1]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -34.0, 95% CI 2-sided [-42.4 to -25.6]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -26.1, 95% CI 2-sided [-34.6 to -17.6]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -21.8, 95% CI 2-sided [-30.3 to -13.3]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -31.5, 95% CI 2-sided [-39.9 to -23.1]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 50 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -29.3, 95% CI 2-sided [-37.3 to -21.4]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -30.8, 95% CI 2-sided [-38.8 to -22.9]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Other; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -39.5, 95% CI 2-sided [-47.4 to -31.6]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -28.9, 95% CI 2-sided [-36.4 to -21.4]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -27.2, 95% CI 2-sided [-34.8 to -19.7]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -34.8, 95% CI 2-sided [-42.3 to -27.4]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -29.2, 95% CI 2-sided [-38.5 to -20.0]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -28.7, 95% CI 2-sided [-37.9 to -19.5]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -36.4, 95% CI 2-sided [-45.5 to -27.2]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -24.3, 95% CI 2-sided [-32.7 to -15.9]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -23.5, 95% CI 2-sided [-31.9 to -15.1]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -31.2, 95% CI 2-sided [-39.5 to -22.9]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -18.6, 95% CI 2-sided [-27.6 to -9.7]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p = 0.0006, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -15.8, 95% CI 2-sided [-24.7 to -6.8]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -22.6, 95% CI 2-sided [-31.4 to -13.8]

5. Secondary Outcome: Percent Change From Baseline in Fasting Total Apolipoprotein B (ApoB) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 46 | 46 | 46 | 48
percentage change | 2.27 (2.807) | -16.40 (2.835) | -12.91 (2.805) | -19.64 (2.788)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -18.66, 95% CI 2-sided [-26.53 to -10.80]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p = 0.0002, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -15.18, 95% CI 2-sided [-23.00 to -7.36]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs. Placebo at Week 24 = -21.90, 95% CI 2-sided [-29.69 to -14.12]

6. Secondary Outcome: Percent Change From Baseline in Fasting Total ApoB Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 50 | 50 | 48 | 49
  Week 4 | 2.57 (2.074) | -14.00 (2.116) | -11.71 (2.093) | -18.47 (2.105)
  Week 8: number analyzed (Participants) | 50 | 50 | 49 | 48
  Week 8 | 1.51 (2.518) | -15.85 (2.553) | -10.66 (2.525) | -15.05 (2.556)
  Week 12: number analyzed (Participants) | 46 | 48 | 48 | 50
  Week 12 | 2.26 (2.656) | -14.96 (2.653) | -7.69 (2.617) | -15.10 (2.606)
  Week 16: number analyzed (Participants) | 48 | 49 | 48 | 50
  Week 16 | -1.36 (2.524) | -15.72 (2.543) | -14.33 (2.513) | -21.66 (2.509)
  Week 20: number analyzed (Participants) | 47 | 48 | 48 | 50
  Week 20 | -0.28 (2.350) | -17.99 (2.370) | -14.52 (2.329) | -18.58 (2.326)
  Week 24: number analyzed (Participants) | 46 | 46 | 46 | 48
  Week 24 | 2.27 (2.807) | -16.40 (2.835) | -12.91 (2.805) | -19.64 (2.788)
  Week 28: number analyzed (Participants) | 47 | 46 | 45 | 48
  Week 28 | 0.51 (2.688) | -15.39 (2.725) | -12.47 (2.703) | -17.03 (2.680)
  Week 36: number analyzed (Participants) | 47 | 47 | 46 | 49
  Week 36 | -2.30 (2.777) | -12.85 (2.801) | -9.07 (2.791) | -13.21 (2.756)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -16.57, 95% CI 2-sided [-22.41 to -10.74]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -14.28, 95% CI 2-sided [-20.08 to -8.48]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -21.04, 95% CI 2-sided [-26.85 to -15.23]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -17.35, 95% CI 2-sided [-24.42 to -10.29]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p = 0.0008, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -12.16, 95% CI 2-sided [-19.19 to -5.13]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -16.56, 95% CI 2-sided [-23.62 to -9.50]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -17.21, 95% CI 2-sided [-24.61 to -9.81]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p = 0.0082, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -9.95, 95% CI 2-sided [-17.30 to -2.60]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -17.35, 95% CI 2-sided [-24.68 to -10.03]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 50 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -14.36, 95% CI 2-sided [-21.42 to -7.30]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p = 0.0003, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -12.97, 95% CI 2-sided [-19.98 to -5.95]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Other; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -20.30, 95% CI 2-sided [-27.30 to -13.29]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -17.71, 95% CI 2-sided [-24.29 to -11.13]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -14.23, 95% CI 2-sided [-20.75 to -7.72]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -18.30, 95% CI 2-sided [-24.80 to -11.79]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -18.66, 95% CI 2-sided [-26.53 to -10.80]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p = 0.0002, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -15.18, 95% CI 2-sided [-23.00 to -7.36]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -21.90, 95% CI 2-sided [-29.69 to -14.12]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -15.90, 95% CI 2-sided [-23.44 to -8.35]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p = 0.0008, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -12.98, 95% CI 2-sided [-20.49 to -5.46]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -17.54, 95% CI 2-sided [-25.01 to -10.07]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p = 0.0081, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -10.55, 95% CI 2-sided [-18.32 to -2.77]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p = 0.0871, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -6.76, 95% CI 2-sided [-14.52 to 0.99]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p = 0.0058, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 2, analysis 1]; Difference = -10.91, 95% CI 2-sided [-18.61 to -3.20]

7. Secondary Outcome: Percent Change From Baseline in Fasting Low-density Lipoprotein-Cholesterol (LDL-C) Using Ultracentrifugation at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 47 | 47 | 47 | 49
percentage change | 5.0 (4.53) | -11.0 (4.58) | -4.3 (4.56) | -15.1 (4.51)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p = 0.0138, Mixed Models Repeated Measures — Model includes treatment arm, study visit, and baseline value as model terms. Model also includes treatment by visit and treatment by baseline as interaction terms; Difference vs. Placebo at Week 24 = -16.0, 95% CI 2-sided [-28.7 to -3.3]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p = 0.1480, Mixed Models Repated Measures — [p-value comment as in outcome 7, analysis 1]; Difference vs Placebo at Week 24 = -9.3, 95% CI 2-sided [-22.0 to 3.3]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p = 0.0019, Mxed Models Repeated Measures — [p-value comment as in outcome 7, analysis 1]; Difference vs Placebo at Week 24 = -20.2, 95% CI 2-sided [-32.8 to -7.5]

8. Secondary Outcome: Percent Change From Baseline in Fasting LDL-C Using Ultracentrifugation Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 51 | 49 | 48 | 50
  Week 4 | 5.1 (3.95) | -8.3 (4.03) | -3.4 (4.02) | -13.7 (3.98)
  Week 8: number analyzed (Participants) | 51 | 50 | 49 | 49
  Week 8 | 3.7 (4.78) | -10.1 (4.85) | -0.7 (4.83) | -10.8 (4.81)
  Week 12: number analyzed (Participants) | 47 | 48 | 48 | 51
  Week 12 | 7.7 (7.31) | -7.6 (7.36) | 7.9 (7.34) | -12.1 (7.23)
  Week 16: number analyzed (Participants) | 49 | 49 | 49 | 51
  Week 16 | 3.6 (4.51) | -9.5 (4.56) | -7.4 (4.52) | -19.5 (4.48)
  Week 20: number analyzed (Participants) | 48 | 48 | 48 | 51
  Week 20 | 1.8 (4.26) | -12.2 (4.31) | -6.9 (4.28) | -15.3 (4.22)
  Week 24: number analyzed (Participants) | 47 | 47 | 47 | 49
  Week 24 | 5.0 (4.53) | -11.0 (4.58) | -4.3 (4.56) | -15.1 (4.51)
  Week 28: number analyzed (Participants) | 48 | 46 | 45 | 49
  Week 28 | 0.2 (4.67) | -9.1 (4.75) | -2.4 (4.74) | -11.3 (4.66)
  Week 36: number analyzed (Participants) | 48 | 47 | 46 | 50
  Week 36 | 3.1 (5.75) | -8.9 (5.81) | 3.7 (5.82) | -4.4 (5.71)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p = 0.0192, Mixed Model Repeated Measures (MMRM) — MMRM model includes treatment arm, study visit, and baseline value as model terms. The model also includes treatment by visit and treatment by baseline as interaction terms; Difference = -13.3, 95% CI 2-sided [-24.5 to -2.2]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p = 0.1362, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -8.4, 95% CI 2-sided [-19.6 to 2.7]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p = 0.0010, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -18.7, 95% CI 2-sided [-29.8 to -7.7]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p = 0.0428, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -13.9, 95% CI 2-sided [-27.3 to -0.5]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p = 0.5122, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -4.5, 95% CI 2-sided [-17.9 to 8.9]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p = 0.0331, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -14.6, 95% CI 2-sided [-27.9 to -1.2]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p = 0.1400, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -15.4, 95% CI 2-sided [-35.8 to 5.1]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p = 0.9854, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = 0.2, 95% CI 2-sided [-20.2 to 20.6]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p = 0.0552, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -19.8, 95% CI 2-sided [-40.1 to 0.4]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 50 mg; Week 16; Test type: Superiority; p = 0.0430, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -13.1, 95% CI 2-sided [-25.7 to -0.4]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p = 0.0871, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -11.0, 95% CI 2-sided [-23.6 to 1.6]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Superiority; p = 0.0004, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -23.1, 95% CI 2-sided [-35.7 to -10.6]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p = 0.0219, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -14.0, 95% CI 2-sided [-25.9 to -2.0]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Superiority; p = 0.1526, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -8.7, 95% CI 2-sided [-20.6 to 3.2]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p = 0.0049, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -17.0, 95% CI 2-sided [-28.9 to -5.2]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p = 0.0138, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -16.0, 95% CI 2-sided [-28.7 to -3.3]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p = 0.1480, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -9.3, 95% CI 2-sided [-22.0 to 3.3]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p = 0.0019, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -20.2, 95% CI 2-sided [-32.8 to -7.5]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p = 0.1660, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -9.3, 95% CI 2-sided [-22.4 to 3.9]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p = 0.6964, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -2.6, 95% CI 2-sided [-15.7 to 10.5]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p = 0.0831, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -11.5, 95% CI 2-sided [-24.5 to 1.5]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p = 0.1425, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -12.0, 95% CI 2-sided [-28.2 to 4.1]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p = 0.9494, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = 0.5, 95% CI 2-sided [-15.6 to 16.6]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p = 0.3535, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 8, analysis 1]; Difference = -7.5, 95% CI 2-sided [-23.5 to 8.4]

9. Secondary Outcome: Percent Change From Baseline in Angiopoietin-like Protein 3 (ANGPTL3) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 47 | 46 | 47 | 49
percentage change | 1.24 (2.801) | -53.02 (2.829) | -68.52 (2.807) | -72.45 (2.761)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p < .0001, mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo = -54.26, 95% CI 2-sided [-62.11 to -46.40]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo at Week 24 = -69.76, 95% CI 2-sided [-77.58 to -61.95]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo at Week 24 = -73.69, 95% CI 2-sided [-81.44 to -65.93]

10. Secondary Outcome: Percent Change From Baseline in ANGPTL3 Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 51 | 49 | 48 | 50
  Week 4 | 5.54 (2.353) | -62.11 (2.388) | -75.25 (2.401) | -79.15 (2.365)
  Week 8: number analyzed (Participants) | 51 | 49 | 49 | 49
  Week 8 | 2.97 (3.023) | -56.09 (3.074) | -69.01 (3.066) | -73.47 (3.045)
  Week 12: number analyzed (Participants) | 47 | 47 | 48 | 51
  Week 12 | 7.38 (3.599) | -47.72 (3.635) | -63.17 (3.608) | -66.62 (3.542)
  Week 16: number analyzed (Participants) | 49 | 48 | 49 | 51
  Week 16 | 8.48 (2.379) | -63.73 (2.400) | -75.61 (2.379) | -80.52 (2.345)
  Week 20: number analyzed (Participants) | 48 | 47 | 48 | 51
  Week 20 | 4.35 (2.338) | -60.50 (2.360) | -73.10 (2.347) | -76.25 (2.299)
  Week 24: number analyzed (Participants) | 47 | 46 | 47 | 49
  Week 24 | 1.24 (2.801) | -53.02 (2.829) | -68.52 (2.807) | -72.45 (2.761)
  Week 28: number analyzed (Participants) | 48 | 46 | 45 | 49
  Week 28 | 5.18 (2.879) | -49.57 (2.920) | -61.43 (2.921) | -68.19 (2.852)
  Week 36: number analyzed (Participants) | 48 | 46 | 46 | 50
  Week 36 | 3.73 (3.110) | -41.70 (3.158) | -53.41 (3.155) | -59.85 (3.066)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — Model includes treatment arm, study visit, randomization stratification factor (level of LDL-C at Screening [≥100 mg/dL versus <100 mg/dL]),and baseline value as model terms. Includes treatment by visit and treatment by baseline as interaction terms; Difference = -67.65, 95% CI 2-sided [-74.26 to -61.04]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -80.80, 95% CI 2-sided [-87.42 to -74.17]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -84.69, 95% CI 2-sided [-91.27 to -78.12]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -59.07, 95% CI 2-sided [-67.57 to -50.57]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -71.98, 95% CI 2-sided [-80.47 to -63.50]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -76.44, 95% CI 2-sided [-84.90 to -67.99]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -55.10, 95% CI 2-sided [-65.18 to -45.01]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -70.55, 95% CI 2-sided [-80.60 to -60.51]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -74.00, 95% CI 2-sided [-83.95 to -64.04]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -72.22, 95% CI 2-sided [-78.88 to -65.56]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -84.09, 95% CI 2-sided [-90.72 to -77.46]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -89.00, 95% CI 2-sided [-95.59 to -82.42]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -64.86, 95% CI 2-sided [-71.40 to -58.31]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -77.45, 95% CI 2-sided [-83.98 to -70.93]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -80.60, 95% CI 2-sided [-87.06 to -74.14]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -54.26, 95% CI 2-sided [-62.11 to -46.40]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -69.76, 95% CI 2-sided [-77.58 to -61.95]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -73.69, 95% CI 2-sided [-81.44 to -65.93]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -54.75, 95% CI 2-sided [-62.84 to -46.67]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -66.60, 95% CI 2-sided [-74.69 to -58.52]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -73.37, 95% CI 2-sided [-81.36 to -65.38]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -45.43, 95% CI 2-sided [-54.17 to -36.69]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -57.15, 95% CI 2-sided [-65.88 to -48.41]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 10, analysis 1]; Difference = -63.58, 95% CI 2-sided [-72.19 to -54.97]

11. Secondary Outcome: Percent Change From Baseline in Fasting High-Density Lipoprotein-Cholesterol (HDL-C) at Week 24
Time Frame: Baseline, Week 24
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 47 | 47 | 47 | 49
percentage change | 3.1 (2.91) | -9.0 (2.94) | -18.5 (2.96) | -21.5 (2.89)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Test type: Superiority; p = 0.0039, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo at Week 24 = -12.0, 95% CI 2-sided [-20.2 to -3.9]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Difference vs Placebo at Week 24 = -21.6, 95% CI 2-sided [-29.8 to -13.4]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Test type: Superiority; p < .0001, Mixed Models Repeated Measures — [p-value comment as in outcome 1, analysis 1]; Differeence vs Placebo at week 24 = -24.5, 95% CI 2-sided [-32.6 to -16.5]

12. Secondary Outcome: Percent Change From Baseline in Fasting HDL-C Over Time
Time Frame: Baseline, up to Week 36 (double-blind treatment period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 51 | 51 | 51
percentage change
  Week 4: number analyzed (Participants) | 51 | 50 | 48 | 50
  Week 4 | -0.3 (2.59) | -13.9 (2.63) | -25.5 (2.68) | -24.8 (2.61)
  Week 8: number analyzed (Participants) | 51 | 50 | 49 | 49
  Week 8 | 0.4 (2.67) | -14.5 (2.71) | -25.0 (2.74) | -25.8 (2.69)
  Week 12: number analyzed (Participants) | 47 | 48 | 48 | 51
  Week 12 | 2.0 (3.10) | -7.0 (3.11) | -18.7 (3.14) | -18.2 (3.05)
  Week 16: number analyzed (Participants) | 49 | 49 | 49 | 51
  Week 16 | 2.1 (2.99) | -15.8 (3.02) | -28.5 (3.04) | -30.2 (2.96)
  Week 20: number analyzed (Participants) | 48 | 48 | 48 | 51
  Week 20 | 3.4 (2.89) | -11.3 (2.92) | -25.1 (2.94) | -27.1 (2.86)
  Week 24: number analyzed (Participants) | 47 | 47 | 47 | 49
  Week 24 | 3.1 (2.91) | -9.0 (2.94) | -18.5 (2.96) | -21.5 (2.89)
  Week 28: number analyzed (Participants) | 48 | 47 | 45 | 49
  Week 28 | 3.0 (2.78) | -5.5 (2.82) | -14.7 (2.87) | -18.6 (2.77)
  Week 36: number analyzed (Participants) | 48 | 47 | 46 | 50
  Week 36 | 6.4 (2.78) | -1.4 (2.82) | -13.7 (2.86) | -9.4 (2.75)
Statistical Analysis 1: Comparison: Placebo vs ARO-ANG3 50 mg; Week 4; Test type: Superiority; p = 0.0003, Mixed Model Repeated Measures (MMRM) — Includes treatment arm, study visit, randomization stratification factor (level of LDL-C at Screening [≥100 mg/dL versus <100 mg/dL]),and baseline value as model terms. Also includes treatment by visit and treatment by baseline as interaction terms; Difference = -13.7, 95% CI 2-sided [-20.9 to -6.4]
Statistical Analysis 2: Comparison: Placebo vs ARO-ANG3 100 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -25.3, 95% CI 2-sided [-32.6 to -17.9]
Statistical Analysis 3: Comparison: Placebo vs ARO-ANG3 200 mg; Week 4; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -24.5, 95% CI 2-sided [-31.8 to -17.3]
Statistical Analysis 4: Comparison: Placebo vs ARO-ANG3 50 mg; Week 8; Test type: Superiority; p = 0.0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -15.0, 95% CI 2-sided [-22.4 to -7.5]
Statistical Analysis 5: Comparison: Placebo vs ARO-ANG3 100 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -25.4, 95% CI 2-sided [-33.0 to -17.9]
Statistical Analysis 6: Comparison: Placebo vs ARO-ANG3 200 mg; Week 8; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -26.2, 95% CI 2-sided [-33.7 to -18.7]
Statistical Analysis 7: Comparison: Placebo vs ARO-ANG3 50 mg; Week 12; Test type: Superiority; p = 0.0429, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -8.9, 95% CI 2-sided [-17.6 to -0.3]
Statistical Analysis 8: Comparison: Placebo vs ARO-ANG3 100 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -20.7, 95% CI 2-sided [-29.4 to -12.0]
Statistical Analysis 9: Comparison: Placebo vs ARO-ANG3 200 mg; Week 12; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -20.1, 95% CI 2-sided [-28.7 to -11.6]
Statistical Analysis 10: Comparison: Placebo vs ARO-ANG3 50 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -17.9, 95% CI 2-sided [-26.2 to -9.5]
Statistical Analysis 11: Comparison: Placebo vs ARO-ANG3 100 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -30.6, 95% CI 2-sided [-39.0 to -22.2]
Statistical Analysis 12: Comparison: Placebo vs ARO-ANG3 200 mg; Week 16; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -32.3, 95% CI 2-sided [-40.5 to -24.0]
Statistical Analysis 13: Comparison: Placebo vs ARO-ANG3 50 mg; Week 20; Test type: Superiority; p = 0.0005, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -14.6, 95% CI 2-sided [-22.7 to -6.5]
Statistical Analysis 14: Comparison: Placebo vs ARO-ANG3 100 mg; Week 20; Test type: Other; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -28.4, 95% CI 2-sided [-36.6 to -20.3]
Statistical Analysis 15: Comparison: Placebo vs ARO-ANG3 200 mg; Week 20; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -30.4, 95% CI 2-sided [-38.4 to -22.4]
Statistical Analysis 16: Comparison: Placebo vs ARO-ANG3 50 mg; Week 24; Test type: Superiority; p = 0.0039, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -12.0, 95% CI 2-sided [-20.2 to -3.9]
Statistical Analysis 17: Comparison: Placebo vs ARO-ANG3 100 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -21.6, 95% CI 2-sided [-29.8 to -13.4]
Statistical Analysis 18: Comparison: Placebo vs ARO-ANG3 200 mg; Week 24; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -24.5, 95% CI 2-sided [-32.6 to -16.5]
Statistical Analysis 19: Comparison: Placebo vs ARO-ANG3 50 mg; Week 28; Test type: Superiority; p = 0.0343, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -8.4, 95% CI 2-sided [-16.2 to -0.6]
Statistical Analysis 20: Comparison: Placebo vs ARO-ANG3 100 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -17.7, 95% CI 2-sided [-25.6 to -9.8]
Statistical Analysis 21: Comparison: Placebo vs ARO-ANG3 200 mg; Week 28; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -21.5, 95% CI 2-sided [-29.3 to -13.8]
Statistical Analysis 22: Comparison: Placebo vs ARO-ANG3 50 mg; Week 36; Test type: Superiority; p = 0.0501, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -7.8, 95% CI 2-sided [-15.6 to 0.0]
Statistical Analysis 23: Comparison: Placebo vs ARO-ANG3 100 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -20.1, 95% CI 2-sided [-27.9 to -12.2]
Statistical Analysis 24: Comparison: Placebo vs ARO-ANG3 200 mg; Week 36; Test type: Superiority; p < .0001, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 12, analysis 1]; Difference = -15.8, 95% CI 2-sided [-23.5 to -8.1]

13. Secondary Outcome: Plasma Pharmacokinetic (PK) Concentration for ARO-ANG3 Over Time in the Double-Blind Treatment Period
Time Frame: Baseline, Day 1: pre-dose, 15 minutes, 1, 3, 6 hours post-dose; Day 2: 24 hours post-dose; Week 12: pre-dose, 15 minutes, 1, 3, 6, 24 hours post-dose (double-blind treatment period)
Population: Full PK Analysis Set: All participants who received at least 1 dose of active study drug and had at least 1 PK concentration data value. Observed cases.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 16 | 21 | 18
ng/mL
  Day 1, Pre-Dose | 0.0000 (0.00000) | 2.6685 (12.22871) | 0.0000 (0.00000)
  Day 1, 15 Minutes Post-Dose | 57.6941 (28.05778) | 63.5267 (55.85108) | 154.7823 (129.43190)
  Day 1, 1 Hour Post-Dose | 75.3752 (31.39048) | 130.3387 (81.73501) | 221.5979 (105.15447)
  Day 1, 3 Hours Post-Dose | 77.9834 (34.90982) | 143.7746 (79.62215) | 259.2799 (144.46149)
  Day 1, 6 Hours Post-Dose | 83.9751 (53.53021) | 152.0097 (91.30854) | 280.0843 (153.62465)
  Day 2, 24 Hours Post-Dose: number analyzed (Participants) | 16 | 20 | 17
  Day 2, 24 Hours Post-Dose | 13.3369 (8.85893) | 33.3047 (16.31049) | 77.9982 (31.94202)
  Week 12, Pre-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, Pre-Dose | 0.0000 (0.00000) | 0.0653 (0.27695) | 1.9366 (7.74650)
  Week 12, 15 Minutes Post-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, 15 Minutes Post-Dose | 54.2741 (43.95835) | 68.3054 (52.28977) | 134.0610 (138.22698)
  Week 12, 1 Hour Post-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, 1 Hour Post-Dose | 76.2131 (34.49650) | 130.2505 (52.66507) | 247.9728 (112.83368)
  Week 12, 3 Hours Post-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, 3 Hours Post-Dose | 78.2496 (36.47898) | 152.0302 (78.31595) | 304.2006 (178.69258)
  Week 12, 6 Hours Post-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, 6 Hours Post-Dose | 87.6919 (37.30155) | 154.3280 (71.93043) | 312.6397 (174.86753)
  Week 12, 24 Hours Post-Dose: number analyzed (Participants) | 14 | 18 | 16
  Week 12, 24 Hours Post-Dose | 15.3604 (13.03807) | 36.2506 (18.33432) | 103.1401 (60.85616)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and/or Serious TEAEs up to Week 24
Description: TEAEs are adverse events (AEs) that occur following IP administration or a pre-existing condition exacerbated following IP administration. An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. A serious adverse event (SAE) is an AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction.
Time Frame: From first dose of IP up to Week 24
Population: Safety Analysis Set: All participants who received at least 1 dose of IP during the study period, analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants
  All TEAEs (Including Serious) | 30 | 37 | 29 | 39
  Serious TEAEs | 3 | 3 | 0 | 1

15. Secondary Outcome: Number of Participants With TEAEs and/or SAEs Over Time in the Double-Blind Treatment Period
Description: Adverse event (AE)=any untoward medical occurrence that does not necessarily have to have a causal relationship with this treatment. TEAEs=AEs with onset after administration of the study drug, or when a pre-existing medical condition increases in severity or frequency after study drug administration. Serious adverse event (SAE)= an AE that results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction.
Time Frame: up to Week 36 (double-blind treatment period)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Pooled): Placebo calculated volume to match active treatment by subcutaneous (sc) injection for Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
Arm/Group | Placebo (Pooled) | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg
Number analyzed (Participants) | 51 | 50 | 51 | 52
Participants
  All Treatment-Emergent Adverse Events (TEAEs) | 35 | 40 | 34 | 42
  Treatment-related TEAEs | 8 | 12 | 8 | 12
  Serious TEAEs | 4 | 5 | 0 | 1
  TEAEs leading to study drug discontinuation | 2 | 0 | 1 | 0
  Deaths | 1 | 0 | 0 | 0
  Local Injection Site Reactions (LISR) | 1 | 0 | 3 | 2

16. Secondary Outcome: Number of Participants With AEs and/or SAEs Over Time in the Open-Label Extension (OLE) Period
Description: as for outcome 15
Time Frame: From first dose of study drug in the OLE up to Month 24 (open-label extension)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Groups:
- Placebo/ARO-ANG3 50mg: Placebo calculated volume to match active treatment by subcutaneous (sc) injection for Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 by sc injection during the open-label extension period.
- ARO-ANG3 50 mg/ARO-ANG3 50 mg: ARO-ANG3 50 mg by sc injection for up to 8 doses during the open-label extension period.
- Placebo/ARO-ANG3 100 mg: Placebo calculated volume to match active treatment ARO-ANG3 100 mg by sc injection for up to 8 doses during the open-label extension period.
- ARO-ANG3 100 mg/ARO-ANG3 100 mg: ARO-ANG3 100 mg by sc injection for up to 8 doses during the open-label extension period.
- Placebo/ARO-ANG3 200 mg: Placebo calculated volume to match active treatment ARO-ANG3 200 mg by sc injection for up to 8 doses during the open-label extension period.
- ARO-ANG3 200 mg/ARO-ANG3 200 mg: ARO-ANG3 200 mg by sc injection for up to 8 doses during the open-label extension period.
Arm/Group | Placebo/ARO-ANG3 50mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200 mg/ARO-ANG3 200 mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
Participants
  All Treatment-Emergent Adverse Events (TEAEs) | 10 | 27 | 13 | 30 | 10 | 31
  Treatment-related TEAEs | 2 | 8 | 4 | 6 | 0 | 6
  Serious TEAEs | 3 | 4 | 2 | 5 | 2 | 5
  TEAEs leading to study drug discontinuation | 0 | 0 | 1 | 2 | 1 | 1
  Deaths | 0 | 0 | 0 | 1 | 0 | 0

17. Secondary Outcome: Percent Change From Baseline in Fasting TG Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Groups:
- Placebo/ARO-ANG3 50 mg: Placebo calculated volume to match active treatment by subcutaneous (sc) injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 50 mg by sc injection during the open-label extension period.
- Placebo/ARO-ANG3 100 mg: Placebo calculated volume to match active treatment by subcutaneous (sc) injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 100 mg by sc injection during the open-label extension period.
Arm/Group | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | -10.02 (8.711) | -34.78 (3.941) | -2.09 (13.925) | -39.64 (3.357) | 7.87 (12.061) | -51.88 (2.612)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 39
  Percent Change from Baseline to OLE Month 1 | -43.74 (5.555) | -45.32 (3.994) | -50.45 (7.323) | -52.86 (3.051) | -49.57 (5.990) | -62.76 (2.262)
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Month 2 | -47.14 (4.687) | -45.78 (4.449) | -48.96 (7.586) | -51.51 (2.712) | -48.98 (6.568) | -58.66 (2.135)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 13 | 36 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 3 | -40.67 (5.792) | -42.51 (3.294) | -42.05 (8.623) | -48.07 (3.255) | -40.73 (8.993) | -56.59 (2.225)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 13 | 36 | 14 | 35 | 12 | 40
  Percent Change from Baseline to OLE Month 6 | -45.81 (7.065) | -48.67 (4.081) | -48.62 (7.597) | -46.81 (3.828) | -46.34 (8.818) | -57.14 (2.697)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 12 | 34 | 12 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 12 | -40.57 (9.384) | -47.10 (3.546) | -52.40 (6.578) | -50.56 (4.288) | -49.06 (3.275) | -58.36 (2.110)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 15 | -47.40 (6.442) | -47.33 (3.969) | -58.81 (4.310) | -56.23 (2.968) | -44.56 (4.440) | -53.57 (4.055)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 18 | -48.07 (6.892) | -48.48 (3.041) | -55.29 (5.170) | -55.11 (3.039) | -49.25 (4.860) | -51.71 (4.761)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 11 | 35 | 10 | 35 | 10 | 36
  Percent Change from Baseline to OLE Month 21 | -41.86 (9.334) | -45.95 (3.609) | -58.42 (3.043) | -55.23 (3.101) | -49.30 (4.388) | -47.42 (6.810)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 5 | 20 | 4 | 20 | 7 | 23
  Percent Change from Baseline to OLE Month 24 | -48.23 (11.315) | -53.83 (3.490) | -61.61 (8.343) | -56.65 (3.545) | -51.88 (3.705) | -58.96 (3.563)

18. Secondary Outcome: Percent Change From Baseline in Fasting Non-HDL-C Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | 6.70 (13.049) | -19.95 (3.532) | -5.02 (5.171) | -16.02 (3.824) | -2.53 (3.750) | -23.12 (3.116)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 39
  Percent Change from Baseline to OLE Month 1 | -14.79 (6.493) | -22.99 (3.544) | -25.80 (4.039) | -25.23 (3.912) | -28.13 (3.930) | -33.41 (3.158)
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Month 2 | -14.70 (5.087) | -25.54 (3.730) | -22.32 (5.340) | -22.98 (3.151) | -28.43 (4.168) | -30.35 (3.013)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 13 | 36 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 3 | -14.32 (6.774) | -20.71 (3.770) | -19.61 (4.659) | -22.97 (3.462) | -25.19 (4.215) | -26.68 (3.107)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 13 | 36 | 14 | 35 | 12 | 40
  Percent Change from Baseline to OLE Month 6 | -10.42 (7.330) | -22.11 (4.372) | -26.53 (4.347) | -24.38 (3.392) | -30.83 (4.832) | -27.84 (3.414)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 12 | 34 | 12 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 12 | -13.72 (9.131) | -22.82 (4.267) | -24.42 (7.159) | -30.48 (3.626) | -28.60 (3.545) | -30.08 (2.731)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 15 | -13.02 (13.661) | -24.01 (4.257) | -25.66 (3.442) | -31.53 (3.040) | -25.86 (4.405) | -27.73 (3.387)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 18 | -23.39 (6.010) | -23.26 (3.579) | -25.34 (4.315) | -33.90 (3.422) | -29.09 (4.005) | -27.88 (3.495)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 11 | 35 | 10 | 35 | 10 | 36
  Percent Change from Baseline to OLE Month 21 | -13.13 (14.219) | -25.07 (3.492) | -34.23 (3.783) | -30.46 (2.642) | -28.66 (4.590) | -25.75 (3.735)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 5 | 20 | 4 | 20 | 7 | 23
  Percent Change from Baseline to OLE Month 24 | -32.24 (14.568) | -27.52 (5.126) | -37.23 (3.633) | -31.95 (4.492) | -24.24 (9.558) | -30.82 (4.407)

19. Secondary Outcome: Percent Change From Baseline in Fasting Total ApoB Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1: number analyzed (Participants) | 12 | 36 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | 6.57 (8.959) | -13.49 (3.086) | -10.22 (4.678) | -7.48 (2.924) | -3.88 (3.080) | -11.77 (3.309)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 1 | 0 | 1 | 1 | 0 | 1
  Percent Change from Baseline to OLE Month 1 | 6.82 (NA) — n=1 |  | -1.65 (NA) — n=1 | -4.45 (NA) — n=1 |  | -21.63 (NA) — n=1
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 4 | 6 | 2 | 6 | 2 | 10
  Percent Change from Baseline to OLE Month 2 | 0.31 (8.213) | -21.00 (6.460) | -3.56 (6.243) | -7.93 (5.968) | -11.37 (16.839) | -7.58 (6.338)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 5 | 13 | 3 | 12 | 4 | 15
  Percent Change from Baseline to OLE Month 3 | -5.48 (13.745) | -13.01 (7.131) | -0.30 (3.518) | -7.09 (5.090) | -13.13 (4.275) | -8.34 (3.722)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 10 | 28 | 11 | 29 | 8 | 31
  Percent Change from Baseline to OLE Month 6 | -1.23 (7.644) | -13.89 (3.645) | -13.84 (3.803) | -11.91 (3.517) | -18.14 (2.810) | -14.04 (3.504)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 11 | 34 | 12 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 12 | -3.46 (9.733) | -12.63 (3.662) | -13.78 (6.382) | -15.14 (3.520) | -13.87 (2.996) | -15.90 (2.835)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 11 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 15 | -8.08 (9.722) | -12.73 (3.587) | -13.40 (3.056) | -16.23 (2.661) | -11.27 (4.524) | -13.05 (3.530)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 11 | 35 | 11 | 35 | 12 | 36
  Percent Change from Baseline to OLE Month 18 | -14.34 (5.296) | -13.83 (3.624) | -14.12 (3.655) | -19.88 (2.991) | -13.63 (3.819) | -13.92 (3.741)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 10 | 35 | 10 | 35 | 10 | 35
  Percent Change from Baseline to OLE Month 21 | 0.08 (10.835) | -13.42 (3.462) | -21.03 (3.791) | -15.03 (2.910) | -15.70 (4.187) | -11.85 (3.789)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 4 | 20 | 4 | 20 | 7 | 22
  Percent Change from Baseline to OLE Month 24 | -6.57 (11.292) | -14.39 (5.371) | -24.76 (4.680) | -16.73 (4.236) | -10.27 (8.790) | -18.04 (4.441)

20. Secondary Outcome: Percent Change From Baseline in Fasting LDL-C Using Ultracentrifugation Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | 16.61 (13.866) | -7.68 (4.934) | -1.59 (8.079) | 4.59 (7.053) | 4.13 (5.905) | -2.82 (5.633)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 39
  Percent Change from Baseline to OLE Month 1 | 6.61 (8.960) | -4.90 (5.203) | -7.43 (5.762) | -0.07 (7.654) | 3.74 (16.591) | -10.01 (4.929)
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Month 2 | 5.75 (6.546) | -10.81 (5.105) | -3.40 (7.119) | 7.38 (12.473) | 3.50 (20.049) | -10.08 (4.989)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 13 | 36 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 3 | 3.79 (8.934) | -2.69 (5.570) | -2.47 (7.839) | 1.94 (7.628) | 5.74 (20.327) | -1.59 (6.358)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 13 | 36 | 14 | 35 | 12 | 40
  Percent Change from Baseline to OLE Month 6 | 16.09 (11.331) | -2.03 (6.503) | -10.68 (5.700) | -9.92 (4.137) | 3.32 (20.431) | -2.80 (6.230)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 12 | 34 | 12 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 12 | 6.95 (14.056) | -2.77 (6.090) | -4.64 (9.376) | -8.25 (7.573) | 4.05 (18.896) | -6.97 (4.466)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 15 | 8.54 (17.305) | -7.84 (6.363) | -6.14 (6.380) | -5.41 (11.638) | 5.82 (18.362) | -7.85 (5.264)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 18 | -9.73 (8.195) | -5.88 (5.801) | -4.52 (7.677) | -13.20 (7.882) | 6.86 (21.962) | -8.43 (5.346)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 11 | 35 | 10 | 35 | 10 | 36
  Percent Change from Baseline to OLE Month 21 | 9.29 (18.925) | -6.14 (5.553) | -12.81 (7.465) | -4.47 (8.744) | -15.64 (7.008) | -2.16 (5.032)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 5 | 20 | 4 | 20 | 7 | 23
  Percent Change from Baseline to OLE Month 24 | -7.17 (22.117) | -10.57 (6.996) | -12.81 (9.496) | -13.83 (5.902) | -9.58 (14.506) | -6.18 (6.423)

21. Secondary Outcome: Percent Change From Baseline in ANGPTL3 Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 41
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | 3.41 (5.372) | -41.57 (4.417) | 4.47 (7.595) | -56.81 (3.166) | 0.79 (4.664) | -59.24 (3.551)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 13 | 34 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 1 | -59.55 (3.490) | -65.83 (2.836) | -77.02 (2.699) | -76.03 (1.982) | -74.62 (3.753) | -77.96 (2.273)
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Month 2 | -53.85 (3.393) | -60.01 (3.812) | -67.75 (4.771) | -71.21 (2.367) | -70.19 (3.928) | -74.59 (2.775)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 13 | 35 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 3 | -43.36 (5.072) | -48.56 (6.842) | -61.65 (4.510) | -65.54 (3.020) | -64.79 (5.478) | -68.91 (3.310)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 12 | 34 | 14 | 35 | 12 | 40
  Percent Change from Baseline to OLE Month 6 | -49.22 (5.280) | -54.18 (4.076) | -67.23 (4.070) | -68.85 (2.867) | -69.38 (3.736) | -67.04 (3.743)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 12 | 33 | 12 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 12 | -55.48 (5.056) | -55.20 (4.666) | -71.03 (4.370) | -69.32 (3.691) | -63.23 (5.801) | -62.00 (4.122)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 12 | 34 | 11 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 15 | -53.01 (3.998) | -52.97 (4.560) | -65.80 (4.669) | -65.28 (6.196) | -64.57 (3.909) | -55.73 (5.734)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 12 | 34 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 18 | -36.82 (9.076) | -39.57 (5.638) | -65.71 (4.877) | -65.97 (3.280) | -61.38 (4.943) | -55.31 (4.725)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 11 | 34 | 10 | 35 | 11 | 36
  Percent Change from Baseline to OLE Month 21 | -40.12 (5.814) | -43.45 (5.176) | -63.26 (4.176) | -64.68 (3.414) | -58.10 (4.837) | -55.43 (4.784)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 5 | 20 | 4 | 20 | 7 | 23
  Percent Change from Baseline to OLE Month 24 | -44.08 (10.028) | -50.18 (6.570) | -48.46 (14.321) | -62.95 (4.439) | -61.52 (3.012) | -63.89 (4.009)

22. Secondary Outcome: Percent Change From Baseline in Fasting HDL-C Over Time in the Open Label Extension (OLE) Period
Time Frame: Baseline, OLE Baseline, Months 1-24 (open-label extension)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200mg
Number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 41
percentage change
  Percent Change from Baseline to OLE Baseline/OLE Day 1 | 13.70 (6.036) | 1.67 (3.360) | 7.70 (5.318) | -12.88 (3.147) | 4.80 (4.562) | -11.26 (3.771)
  Percent Change from Baseline to OLE Month 1: number analyzed (Participants) | 13 | 35 | 14 | 39 | 13 | 39
  Percent Change from Baseline to OLE Month 1 | -10.68 (8.416) | -12.31 (3.791) | -26.62 (4.804) | -28.81 (3.214) | -14.33 (8.371) | -28.27 (3.705)
  Percent Change from Baseline to OLE Month 2: number analyzed (Participants) | 13 | 36 | 14 | 39 | 13 | 40
  Percent Change from Baseline to OLE Month 2 | -9.46 (6.308) | -10.98 (3.588) | -19.64 (4.846) | -24.78 (3.397) | -13.48 (7.252) | -28.24 (3.362)
  Percent Change from Baseline to OLE Month 3: number analyzed (Participants) | 13 | 36 | 14 | 38 | 13 | 38
  Percent Change from Baseline to OLE Month 3 | -8.80 (5.376) | -9.96 (3.318) | -15.50 (4.847) | -22.29 (3.771) | -12.81 (5.209) | -19.78 (3.504)
  Percent Change from Baseline to OLE Month 6: number analyzed (Participants) | 13 | 36 | 14 | 35 | 12 | 40
  Percent Change from Baseline to OLE Month 6 | -8.26 (6.279) | -3.95 (4.247) | -21.38 (6.028) | -26.54 (3.486) | -13.75 (6.207) | -20.43 (4.082)
  Percent Change from Baseline to OLE Month 12: number analyzed (Participants) | 12 | 34 | 12 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 12 | -13.83 (7.363) | -16.58 (3.672) | -22.23 (5.893) | -26.51 (3.816) | -5.47 (5.504) | -18.32 (4.314)
  Percent Change from Baseline to OLE Month 15: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 38
  Percent Change from Baseline to OLE Month 15 | -9.01 (6.448) | -12.02 (5.116) | -19.76 (5.356) | -29.44 (3.110) | -14.07 (5.004) | -15.04 (4.116)
  Percent Change from Baseline to OLE Month 18: number analyzed (Participants) | 12 | 35 | 11 | 35 | 12 | 37
  Percent Change from Baseline to OLE Month 18 | -10.53 (6.499) | -4.80 (5.980) | -21.60 (5.268) | -28.55 (3.462) | -11.86 (4.787) | -16.39 (4.648)
  Percent Change from Baseline to OLE Month 21: number analyzed (Participants) | 11 | 35 | 10 | 35 | 10 | 36
  Percent Change from Baseline to OLE Month 21 | -3.87 (6.823) | -12.48 (3.816) | -22.77 (4.713) | -26.12 (3.535) | -16.68 (2.024) | -17.82 (3.788)
  Percent Change from Baseline to OLE Month 24: number analyzed (Participants) | 5 | 20 | 4 | 20 | 7 | 23
  Percent Change from Baseline to OLE Month 24 | -8.97 (10.168) | -11.66 (5.293) | -20.28 (15.397) | -27.31 (4.225) | -16.01 (3.759) | -24.10 (5.009)

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization through Month 24. Adverse events: From first dose of study drug through Week 36 (double-blind period); from first dose of open-label study drug up to Month 24 (open-label extension).
Description: Safety Analysis Set: All participants who received at least 1 dose of IP during the study period, analyzed according to the treatment they actually received.
Groups:
- Placebo: Placebo calculated volume to match active treatment by subcutaneous (sc) injection at Day 1 and Week 12 during the double-blind treatment period.
- ARO-ANG3 50 mg: ARO-ANG3 50 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period.
- ARO-ANG3 100 mg: ARO-ANG3 100 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period.
- ARO-ANG3 200 mg: ARO-ANG3 200 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period.
- ARO-ANG3 200mg/ARO-ANG3 200 mg: ARO-ANG3 200 mg by sc injection at Day 1 and Week 12 during the double-blind treatment period. Up to 8 doses of ARO-ANG3 200 mg by sc injection during the open-label extension period.
Arm/Group | Placebo | ARO-ANG3 50 mg | ARO-ANG3 100 mg | ARO-ANG3 200 mg | Placebo/ARO-ANG3 50 mg | ARO-ANG3 50 mg/ARO-ANG3 50 mg | Placebo/ARO-ANG3 100 mg | ARO-ANG3 100 mg/ARO-ANG3 100 mg | Placebo/ARO-ANG3 200 mg | ARO-ANG3 200mg/ARO-ANG3 200 mg
All-Cause Mortality (participants affected / at risk) | 1/51 | 0/50 | 0/51 | 0/52 | 0/13 | 0/36 | 0/14 | 1/39 | 0/13 | 0/41
Serious Adverse Events (participants affected / at risk) | 4/51 | 5/50 | 0/51 | 1/52 | 3/13 | 4/36 | 2/14 | 5/39 | 2/13 | 5/41
Other Adverse Events (participants affected / at risk) | 41/51 | 38/50 | 41/51 | 42/52 | 10/13 | 31/36 | 14/14 | 34/39 | 11/13 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | ARO-ANG3 50 mg (N=50) | ARO-ANG3 100 mg (N=51) | ARO-ANG3 200 mg (N=52) | Placebo/ARO-ANG3 50 mg (N=13) | ARO-ANG3 50 mg/ARO-ANG3 50 mg (N=36) | Placebo/ARO-ANG3 100 mg (N=14) | ARO-ANG3 100 mg/ARO-ANG3 100 mg (N=39) | Placebo/ARO-ANG3 200 mg (N=13) | ARO-ANG3 200mg/ARO-ANG3 200 mg (N=41)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Silent myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic ketosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=51) | ARO-ANG3 50 mg (N=50) | ARO-ANG3 100 mg (N=51) | ARO-ANG3 200 mg (N=52) | Placebo/ARO-ANG3 50 mg (N=13) | ARO-ANG3 50 mg/ARO-ANG3 50 mg (N=36) | Placebo/ARO-ANG3 100 mg (N=14) | ARO-ANG3 100 mg/ARO-ANG3 100 mg (N=39) | Placebo/ARO-ANG3 200 mg (N=13) | ARO-ANG3 200mg/ARO-ANG3 200 mg (N=41)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Splenic cyst (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic valve sclerosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Heart failure with reduced ejection fraction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Suprventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Chalazion (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 4 | 4 | 0 | 1 | 1 | 4 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 3 | 1 | 2 | 0 | 2 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Administration site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 2 | 1 | 0 | 1 | 2 | 2 | 1 | 1
Influenza like illness (General disorders) | 3 | 2 | 3 | 1 | 1 | 2 | 1 | 3 | 1 | 1
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 0 | 2 | 6 | 1 | 0 | 0 | 2 | 0 | 6
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 5 | 7 | 3 | 0 | 4 | 0 | 6 | 0 | 2
Injection site pruritus (General disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 3 | 1 | 0 | 3 | 1 | 3 | 0 | 1
Peripheral swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 3 | 4 | 2 | 0 | 2 | 1 | 4 | 0 | 2
COVID-19 (Infections and infestations) | 14 | 16 | 16 | 18 | 3 | 14 | 5 | 13 | 4 | 15
Conjunctivitis (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 0 | 1 | 2 | 0 | 0 | 3 | 1 | 0 | 2
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infective exacerbation of asthma (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 0 | 3
Labyrinthitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pyuria (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 4 | 3 | 0 | 4 | 1 | 3 | 2 | 0 | 1 | 4
Subcutaneous abscess (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 8 | 9 | 11 | 1 | 6 | 3 | 9 | 2 | 9
Urinary tract infection (Infections and infestations) | 5 | 6 | 6 | 12 | 2 | 4 | 2 | 4 | 1 | 8
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Wound infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 3 | 0 | 1 | 2 | 2 | 3 | 0 | 0
Ear canal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 1 | 3 | 1 | 0 | 2 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 0 | 3
Blood potassium decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 2 | 4 | 3 | 0 | 0 | 4 | 2 | 3 | 0 | 0
High density lipoprotein decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 3 | 3 | 0 | 1 | 0 | 2 | 0 | 3
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4 | 2 | 7 | 0 | 3 | 3 | 2 | 1 | 7
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4 | 4 | 0 | 3 | 3 | 4 | 1 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 8 | 0 | 5 | 0 | 2 | 1 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 0 | 1 | 0 | 2 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4 | 0 | 2 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 3 | 0 | 1 | 1 | 3 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3 | 5 | 1 | 2 | 0 | 3 | 0 | 5
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 4 | 1 | 0 | 2 | 0 | 2 | 1 | 1
Headache (Nervous system disorders) | 6 | 6 | 3 | 9 | 1 | 4 | 3 | 3 | 1 | 6
Hypokinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Renal cyst (Renal and urinary disorders) | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4 | 0 | 3 | 1 | 0 | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 1
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 2 | 5 | 0 | 2 | 0 | 2 | 1 | 4
Superficial vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor retains first right to publish results for this multi-center study, and thereafter can review results communications prior to release and can embargo communications regarding trial results for a period that is 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication of results but can require removal of its confidential information (excluding results).

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/71/NCT04832971/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT04832971/SAP_001.pdf